CLINICAL TRIAL: NCT04465019
Title: The Use of the Exoskeleton Robotic Device in the Rehabilitation of Traumatic Brain Injury
Brief Title: Exoskeleton Rehabilitation on TBI
Acronym: Ekso-TBI
Status: Completed | Type: Observational
Sponsor: DHR Health Institute for Research and Development (Other)
Responsible Party: Principal Investigator, Lisa Trevino, Vice President, DHR Health Institute for Research and Development
Other Study IDs: 1492252
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Traumatic Brain Injury; Cerebral Stroke
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- TBI Group: Subjects in the TBI group included patients who suffered a TBI and who used the EKSO® bionic exoskeleton during their rehabilitation treatment from 01/01/2017 to 04/30/2020.
  Interventions: Device: Exoskeleton Rehabilitation
- CVA Group: Subjects in the CVA group included all patients in the hospital that used the EKSO® during their rehabilitation process during their rehabilitation treatment from 01/01/2017 to 04/30/2020.
  Interventions: Device: Exoskeleton Rehabilitation

INTERVENTIONS:
Device: Exoskeleton Rehabilitation — The EKSO GT® was operated by a Licensed Physical Therapist who was certified to control the device. We followed a strictly established protocol for operating the device during the rehabilitation process as established by the company.

SUMMARY:
Background: Traumatic brain injury (TBI) is one of the leading causes of disability in the United States. The EKSO GT Bionics® (EKSO®) is a robotic exoskeleton approved by the Federal Drug Administration (FDA) for rehabilitation following a cerebrovascular accident (CVA or stroke) and recently received approval for use in patients with TBI. The aim of the study was to examine if the use of exoskeleton rehabilitation in patients with TBI will produce beneficial outcomes. Methods: This retrospective chart-review reports the use of the (EKSO®) robotic device in the rehabilitation of patients with TBI compared to patients with CVA. The investigators utilized data from a single, private rehabilitation hospital for patients that received post-CVA or post-TBI robotic exoskeleton intervention. All patients that used the exoskeleton were discharged from the hospital between 01/01/2017 to 04/30/2020. Ninety-four percent (94%) of patients in the CVA groups and 100% of patients in the TBI group were of Hispanic or Latino ethnicity. Gains in total Functional Independence Measure (FIM), walking and cognition, and length of stay in the rehabilitation facility were measured. Results: Patients in the TBI group (n=11) were significantly younger than the patients in the CVA group (n=66; p< 0.05). Both groups spent a similar amount of time active, number of steps taken, and the number of sessions in the exoskeleton. Both groups also started with similar admission FIM scores. The FIM gain in the TBI group was similar to that of the CVA group (37.5 and 32.0 respectively). The length of stay between groups was not different either. Conclusions: The use of exoskeleton rehabilitation in patients with TBI appear to produce similar outcomes as for patients with CVA, prompting further attention of this intervention for this type of injury.

DETAILED DESCRIPTION:
Study Design and Setting

This is an observational, retrospective, chart review cohort study of patients from a private single rehabilitation hospital. Study approval was granted by the local Institutional Review Board and conformed to the Declaration of Helsinki and the US Federal Policy for the Protection of Human Subjects. Due to the retrospective nature of the study, a full waiver of authorization under the Health Insurance Portability and Accountability Act (1996) was submitted by the study team and approved by the Institutional Review Board.

Participants

Inclusion and Exclusion criteria: Subjects in the TBI group included patients who suffered a TBI and who used the EKSO® bionic exoskeleton during their rehabilitation treatment from 01/01/2017 to 04/30/2020. Subjects in the CVA group included all patients in the hospital that used the EKSO® during their rehabilitation process during the same period of the patients in the TBI group. Patients were excluded if their injury type was outside the scope of the current study. The registered nurse at the rehabilitation facility identified the patients based on the inclusion criteria, and this was verified by the doctor in physical therapy who oversees the rehabilitation hospital patient population. Approval and implementation of the EKSO® bionic device at the hospital commenced in 2014 for patients that suffered a CVA and spinal cord injury. Main indications for the use of the EKSO® during rehabilitation included a height range between 1.56 to 1.9 meters and a patient's weight equal to or less than 100kg. Stable blood pressure was required, with the ability to follow one to two steps commands, and the patient should also have demonstrated a normal range of motion in hips, knees, and ankles.

Variables

Demographic factors considered in this study were age at the time of admission into the rehabilitation facility (measured in years), and patient's sex (males or females). Ethnicity was self-reported and collected in the study, but it was not considered as a covariate since the vast majority of our cohort was of Hispanic origin. The overrepresentation of Hispanics/Latinos in the current cohort responds to the demographic distribution of the area the hospital serves. The investigators collected information related to the impairment type produced by the CVA, and for the TBI; investigators collected the abbreviated injury scale (ASI) to determine the injury severity score (ISS).

The change in FIM score from admission to discharge was used as the primary outcome for this study. The FIM score evaluates the ability of the patient in day-to-day functions within three (3) major categories: self-care, mobility, and communication. To explore whether the use of EKSO® facilitates the improvement in mobility and communication, investigators also explored the motor FIM and social interaction FIM, problem-solving FIM, and memory FIM. In parallel to FIM, investigators evaluated how the length of stay in the facility affected the outcomes.

Data sources/measurements

Variables collected in this study were retrospectively obtained from the patient's electronic medical chart. All information presented in this study was part of the patient's standard of care. No additional intervention or data collection instrument was implemented. The standard of care of the patient is as follows: all potentially eligible candidates were identified and cleared by the physician with subsequent patient education regarding the use of the EKSO®. For the use of the exoskeleton during the rehabilitation process, signed informed consent was obtained from either the patient or designated family member, depending on the status of the patient. Data obtained during the active use of the exoskeleton was visualized in the screen of the EKSO® (time active, steps taken, etc.) and subsequently recorded in each patient's paper chart. This paper was then scanned and uploaded into the patient's electronic chart under his/her progress notes. The therapy technicians helped in the data recording process. All available data related to EKSO use for CVA and TBI at our facility were included in the current study. The primary goal of the data analysis was to gather preliminary comparative outcomes that could guide us into designing larger-controlled studies.

Reduction of Bias

To minimize selection bias in the current study, investigators used all patients that were clinically determined by the attending physician to meet the criteria for exoskeleton rehabilitation. Patients were included in the chart review regardless of the number of sessions of exoskeleton use. All therapist and nurses at our facility have been certified to use the FIM assessment tool and the data is entered using the Uniform Data System for Medical Rehabilitation (https://www.udsmr.org/) software integrated within the hospital medical record platform. The main data extractor in the study (A.M.) is the site expert for data management within the Uniform Data System. Quality of the data was verified by the lead doctor in Physical Therapy (M.E.A.). None of the patients that used exoskeleton in rehabilitation had missing data during the time period used for the current study and all patients in the cohort completed the recommended therapeutic program and were successfully discharged from the hospital.

Exoskeleton use protocol

The EKSO GT® was operated by a Licensed Physical Therapist who was certified to control the device. The device is only approved to be used in a clinical setting. For the purposes of this study, four different modes were utilized to engage and challenge the patients: Pre-Gait, First Step, Pro Step Plus, and 2 Free. Pre-Gait Mode focused on the following metrics to facilitate movement and active participation: bilateral weight shifting in standing with biofeedback, mini squats, and stationary unilateral lower extremity advancement. The First Step mode allowed the therapist to be in full control of all movement. The therapist triggered the initiation and execution of each step reciprocally with the push of a button. In the Pro Step Plus mode, there was an appropriate weight shift either done independently by the patient or facilitated by the therapeutic handling of the physical therapist. The patient was given the opportunity to initiate each step; the EKSO® device completed any incomplete steps. The most advanced mode is called 2 Free. This mode was used to challenge the patient across the continuum as they progress. The patient was responsible for initiating and executing each step. The therapist programmed resistance unilaterally or bilaterally to the lower extremities to increase the demand for the activity.

Statistical methods

Descriptive statistics for the entire study population were generated. Normally distributed continuous variables were described with means and standard deviations, medians and ranges were used for non-normally distributed variables, and frequencies and column percentages summarized categorical variables. Differences in demographic and clinical characteristics between the two treatment groups were evaluated using Student t-test for independent samples for normally distributed continuous variables, Mann-Whitney U test for non-normally distributed continuous variables, and Fisher exact test for categorical variables. To test for the difference between the CVA and TBI groups in respect to socio-demographic and treatment measurements, paired t-test or Wilcoxon signed-rank test for continuous variables and Chi-square test/Fisher exact test for categorical variables were used. Shapiro-Wilk test for normality was conducted to determine the normality of the continuous variables' distributions. Linear regression analyses were carried out to evaluate the associations of each of the outcome variables with age, sex, and length of hospital stay, and with the injury groups (CVA and TBI) variable. All statistical tests were two-sided and were performed at a significance level of 0.05. All statistical analyses were conducted using SAS 9.4 (SAS Institute, Inc, Cary, North Carolina, USA.).

ELIGIBILITY:
Inclusion Criteria:

* Main indications for the use of the EKSO® during rehabilitation included a height range between 1.56 to 1.9 meters and a patient's weight equal to or less than 100kg.
* Stable blood pressure was required, with the ability to follow one to two steps commands, and the patient should also have demonstrated a normal range of motion in hips, knees, and ankles.
* Patient must have suffered a traumatic brain injury or stroke

Exclusion Criteria:

* Patients were excluded if their injury type was outside the scope of the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 66 (10.7%) and 11 (7.9%) patients met the criteria and agreed to use the exoskeleton for CVA and TBI respectively. More than 90% of the study population is of Hispanic ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Functional Independence Measure | Ten weeks
  Increase in FIM from Admission to Discharge

SECONDARY OUTCOMES:
Number of steps taken in the exoskeleton | Inpatient stay at the rehabilitation hospital
Time active in the exoskeleton | Inpatient stay at the rehabilitation hospital

CONTACTS AND LOCATIONS:
Locations (1):
- DHR Health Rehabilitation Hospital, Edinburg, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Interested parties must contact the corresponding author to provide individual data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Up to two years after data publication
Access Criteria: Contact Principal Investigator

REFERENCES:
- [Derived] Trevino LR, Roberge P, Auer ME, Morales A, Torres-Reveron A. Predictors of Functional Outcome in a Cohort of Hispanic Patients Using Exoskeleton Rehabilitation for Cerebrovascular Accidents and Traumatic Brain Injury. Front Neurorobot. 2021 Jun 10;15:682156. doi: 10.3389/fnbot.2021.682156. eCollection 2021. PMID 34177511